CLINICAL TRIAL: NCT02298868
Title: Safety and Efficacy of Baclofen for Treatment of Muscle Spasms in Patients With Cirrhosis: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Zachary Henry, MD, Fellow Physician, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16306
Record Dates: First submitted 2014-11-12; First posted 2014-11-24 (Estimated); Results first posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Muscle Cramps; Cirrhosis
MeSH Terms: conditions — Muscle Cramp; Fibrosis | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): All patients will be administered a standing dose of Baclofen initially at 5 mg three times a day for the first week and then increased to 10 mg three times a day for the next 3 weeks with a tapering dose the final week, a total of 5 weeks of therapy.
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the medication Baclofen for treatment of muscle cramps in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* Presence of muscle cramps on a regular basis

Exclusion Criteria:

* Allergy or hypersensitivity to Baclofen
* Active or untreated Portosystemic encephalopathy
* Active alcohol or substance abuse
* Age less than 18
* Pregnancy
* Concomitant use of narcotic pain medication, other muscle relaxer, or other anti-spastic agent
* Concomitant use of Tricyclic Antidepressant due to drug interaction
* History of chronic kidney disease defined by GFR < 30 (using MDRD equation)
* Subject is institutionalized or a prisoner
* Inability or unwillingness to give informed consent
* Expected lifespan less than 3 months
* Severe or poorly controlled coexisting medical conditions or other significant issues as determined by the principal investigator to hinder the ability to adhere to study protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Henry, M.D., Principal Investigator — University of Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 10
Completed | 7
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Patient underwent transplant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability (Headache)
Description: Proportion of patients with headache at any time during the 4 weeks of therapy
Time Frame: 4 weeks of active therapy
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 10
participants | 3

2. Secondary Outcome: Efficacy of Baclofen to Change Frequency of Muscle Cramps in Patients With Cirrhosis at the End of 4 Weeks of Therapy
Description: Patients undertook a muscle cramp questionnaire prior to treatment that measured frequency in the number of days in a week that a subject experienced muscle cramps. This measures was repeated after 4 weeks of therapy and reported as the mean decrease in frequency of muscle cramps (4 weeks of therapy-Baseline).
Time Frame: Baseline to 4 weeks of therapy
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Treatment
Number analyzed (Participants) | 10
days/week | -4.4 (3.3)

3. Secondary Outcome: Efficacy of Baclofen to Change Severity of Muscle Cramps in Patients With Cirrhosis After 4 Weeks of Therapy
Description: Patients undertook a muscle cramp questionnaire prior to treatment that measured severity in a 0-10 analog scale (0 is no pain and 10 is most severe pain). These measures were repeated after 4 weeks of therapy and the difference was assessed (4 weeks of therapy-Baseline).
Time Frame: Baseline to end of 4 weeks of therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
units on a scale | -6 (2.9)

4. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability (Nausea)
Description: Proportion of patients with nausea at any time during the 4 weeks of therapy
Time Frame: 4 weeks of active therapy
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 10
participants | 4

5. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability (Dizziness)
Description: Proportion of patients with dizziness at any time during the 4 weeks of therapy
Time Frame: 4 weeks of active therapy
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 10
participants | 2

6. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability (Encephalopathy)
Description: Proportion of patients with endephalopathy at any time during the 4 weeks of therapy
Time Frame: 4 weeks of active therapy
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 10
participants | 0

7. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability (Somnolence)
Description: Proportion of patients with somnolence at any time during the 4 weeks of therapy
Time Frame: 4 weeks of active therapy
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 10
participants | 1

8. Secondary Outcome: Change in Frequency of Muscle Cramps After Washout Period
Description: Subjects undertook a muscle cramp questionnaire prior to treatment that measured frequency in the number of days in a week that a subject experienced muscle cramps and repeated this measure at the end of baclofen therapy (end of week 4). Subjects then underwent a 1 week taper of baclofen and a subsequent two week washout period. At the end of the washout period (end of week 7) the subjects underwent a final muscle cramp questionnaire to reassess frequency of muscle cramps. This was then compared to the end of therapy frequency to document the increase in muscle cramps after stopping baclofen. (week 7 result - week 4 result)
Time Frame: End of treatment (week 4) to end of washout (week 7)
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Treatment
Number analyzed (Participants) | 10
days/week | 3.0 (3.9)

9. Secondary Outcome: Change in Severity of Muscle Cramps After Washout Period
Description: Subjects undertook a muscle cramp questionnaire prior to treatment that measured severity on a 0-10 analog scale (0 is no pain, 10 is most severe pain) and repeated this measure at the end of baclofen therapy (end of week 4). Subjects then underwent a 1 week taper of baclofen and a subsequent two week washout period. At the end of the washout period (end of week 7) the subjects underwent a final muscle cramp questionnaire to reassess severity of muscle cramps. This was then compared to the end of therapy severity to document the increase in muscle cramps after stopping baclofen. (week 7 result - week 4 result)
Time Frame: End of treatment (week 4) to end of washout (week 7)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
units on a scale | 4.0 (4.0)

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=10)
Headache (Nervous system disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes